CLINICAL TRIAL: NCT01385293
Title: Phase II Study of BKM120 in Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: BKM120 in Metastatic Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped at the first stage due to futility
Sponsor: Andrew J. Armstrong, MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Andrew J. Armstrong, MD, Assoc Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00027410
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer; Metastatic (Spread to Other Areas of the Body)
Keywords: BKM120; prostate cancer; metastatic castrate-resistant prostate cancer (mCRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): BKM120 at 100mg orally daily
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — BKM120 at the maximum tolerated dose (MTD) of 100mg orally daily
  Other Names: BKM-120

SUMMARY:
The purpose of this study is to evaluate the effects of the study drug, BKM120. The study drug, BKM120, is an inhibitor of a protein called phosphatidyl inositol-3-kinase (PI3K). This protein is found in normal cells and in cancer cells, but often in many cancer cells this protein is overactive. Inhibiting the protein may slow the growth of prostate cancer but this has not been tested yet in men with prostate cancer.

DETAILED DESCRIPTION:
This is an open label, single arm phase II study of BKM120 in men with metastatic castration resistant prostate cancer (CRPC) who have progressed on or following completion of docetaxel-based chemotherapy. Prior progression on cabazitaxel, provenge, abiraterone, or enzalutamide (MDV3100) is also permitted. Patients must have baseline evaluations performed prior to the first dose of study drug and must meet all inclusion and exclusion criteria. Results of the baseline evaluations, which assure that all inclusion and exclusion criteria have been satisfied, must be reviewed by the Principal Investigator or his/her designee prior to enrollment of that patient. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent must be obtained from the patient prior to protocol-specific screening tests. The following criteria apply to all patients enrolled onto the study unless otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky performance status ≥ 70
* Life expectancy of ≥ 12 weeks as determined by treating investigator
* Adequate laboratory parameters
* Histologically confirmed diagnosis of adenocarcinoma of the prostate. Histologic variants of prostate cancer, including neuroendocrine features and small cell carcinoma of the prostate are permitted
* Radiographic evidence of metastatic disease
* Evidence of disease progression on androgen deprivation therapy (ADT)
* A minimum of 4 weeks elapsed off of antiandrogen therapy prior to registration (i.e. flutamide, nilutamide) and 6 weeks for bicalutamide, without evidence of an anti-androgen withdrawal response. Patients who did not have a PSA decline with the most recent antiandrogen therapy require only a 2 week washout period prior to registration
* A minimum of 2 weeks from prior abiraterone acetate, sipuleucel-T, MDV3100, orteronel (TAK700), ketoconazole, or other experimental anti-cancer therapies prior to registration is required. Concomitant treatment with enzalutamide is permitted.
* At least one prior systemic chemotherapy regimen FDA approved for metastatic prostate cancer
* A minimum of 4 weeks from any major surgery prior to registration

Exclusion Criteria:

* Have received prior treatment with a PI3K inhibitor
* Known hypersensitivity to BKM120 or to its excipients
* Untreated brain metastases
* Patients with hepatitis B or C, other acute or chronic liver disease, or a recent (within 12 months of administration of first dose of study drug) history of pancreatitis
* Patients with certain mood disorders as judged by the investigator or a psychiatrist
* History of treatment in an inpatient psychiatric setting
* Concurrent severe and/or uncontrolled cardiac conditions which could compromise participation in the study
* Other concurrent severe and/or uncontrolled concomitant medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol
* Uncontrolled diabetes mellitus defined as a fasting plasma glucose level of >120.
* Diarrhea ≥ CTCAE grade 2
* Drugs or substances known to be strong inhibitors or inducers of the isoenzyme CYP3A4 should be avoided as systemic therapy in association with BKM120 as these can alter its metabolism. Topical use of creams or other applications not absorbed into the circulation is permitted
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Have been treated with any granulocyte colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Currently receiving treatment with medication that has the potential to significantly prolong the QT interval or induce Torsades de Pointes, and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Have received immunosuppressive therapy including corticosteroids ≤ 2 weeks prior to starting study drug. Prednisone at a total daily dose of 10 mg orally or its equivalent is permitted, if initiated at least 2 weeks prior to enrollment
* History of solid organ or stem cell transplantation
* Have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy prior to administration of first dose of study drug
* Have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy prior to administration of first dose of study drug
* Currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell or squamous cell carcinoma of the skin or low grade papillary bladder cancer Other inclusion and exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, ScM, Principal Investigator — Duke Cancer Institute
Locations (3):
- United States (3):
  - Duke Cancer Institute, Durham, North Carolina
  - OHSU Knight Cancer Institute, Portland, Oregon
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- BKM 120: BKM120 at 100mg orally daily
Period: Overall Study
Arm/Group | BKM 120
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BKM 120
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 67 [48 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Prostate Cancer Working Group 2 (PCWG2) Criteria or Based on the Onset of a Skeletal Related Event.
Description: Time in months from the start of study treatment to the date of first progression or death due to any cause. Progression was determined either radiographically using a composite of the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and Prostate Cancer Working Group 2 (PCWG2) criteria or clinically as judged from a skeletal-related event, need for change in therapy, or clinical deterioration. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
  Response and progression are evaluated using a combination of Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and guidelines for prostate cancer endpoints developed by the Prostate Cancer Clinical Trials Working Group (PCWG2). Per RECIST, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM 120
Number analyzed (Participants) | 30
months | 1.9 [1.7 to 3.0]

2. Secondary Outcome: Radiologic Response
Description: The number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. Response and progression is evaluated using a combination of the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) and the guidelines for prostate cancer endpoints developed by the Prostate Cancer Clinical Trials Working Group (PCWG2). Per RECIST, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | BKM 120
Number analyzed (Participants) | 30
participants | 0

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of patients experiencing grade 3-5 adverse events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 28 days post last study drug dose. This is the follow-up safety visit.
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | BKM 120
Number analyzed (Participants) | 30
participants | 16

4. Secondary Outcome: Prostate Specific Antigen (PSA) Response
Description: The number of patients with a 30% and 50% decrease in PSA from baseline.
Time Frame: 2 years
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | BKM 120
Number analyzed (Participants) | 30
participants
  30% Decrease | 1
  50% Decrease | 0

5. Secondary Outcome: Overall Survival of Participants.
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 5 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM 120
Number analyzed (Participants) | 30
months | 10.6 [6.5 to 14.6]

6. Secondary Outcome: Change in Circulating Tumor Cell (CTC) Levels From Baseline
Description: The number of patients with a baseline CTC level of at least 5 who achieved a CTC level of less than 5 during the study.
Time Frame: 2 years
Population: 13 patients had measured CTC levels above 5 at baseline
Measure: Number; unit: participants
Arm/Group | BKM 120
Number analyzed (Participants) | 13
participants | 1

7. Secondary Outcome: Time to New Metastatic Disease From the Baseline Visit
Description: Time in days from the start of study treatment to time of new metastatic disease. Time to new metastatic disease is, defined from the date of first study agent administration to the onset of a new evaluable site of disease as per PCWG2 and RECIST 1.1 guidelines, excluding the primary site and all sites documented at baseline will be assessed. Only those patients that experienced a new lesion per this definition are included.
Time Frame: 5 years
Population: Only those patients that experienced a new lesion per this definition are included.
Measure: Median (Full Range); unit: days
Arm/Group | BKM 120
Number analyzed (Participants) | 12
days | 55 [38 to 108]

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from the start of treatment through the end Up to 28 days post last study drug dose. This is the follow-up safety visit.
Arm/Group | BKM 120
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM 120 (N=30)
Hypotension (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Bronchial Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Pain, worsening bone (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Acute Renal Failure (Renal and urinary disorders) | 1
Urethral obstruction (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM 120 (N=30)
Anemia (Blood and lymphatic system disorders) | 5
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Eye disorder, other (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal pain, right side (Gastrointestinal disorders) | 1
Bloat (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Epigastric pain (Gastrointestinal disorders) | 1
GI virus (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Lip pain (dry lips) (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 10
Stomach pain (Gastrointestinal disorders) | 2
Stomatitis/mouth ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 13
Gait Unsteadiness/imbalance (General disorders) | 1
Generalized cold sensation (General disorders) | 1
Left shoulder pain (General disorders) | 1
Right rib pain (General disorders) | 1
Liver Dysfunction (Hepatobiliary disorders) | 1
Flu virus (Infections and infestations) | 1
Fungal infection, tongue (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Abrasions (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Sunburn (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Creatinine increased (Investigations) | 4
Investigation (Investigations) | 1
Lipase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Serum amylase increased (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and Nutrition (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (spasmatic pain) (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pain, Bilateral rib/flank (Musculoskeletal and connective tissue disorders) | 1
Pain, jaw (Musculoskeletal and connective tissue disorders) | 1
Pain, mid back to ribs (Musculoskeletal and connective tissue disorders) | 1
Pain, worsening bone (Musculoskeletal and connective tissue disorders) | 1
Pain- mid spine, shoulder (Musculoskeletal and connective tissue disorders) | 1
Pain- right femur (Musculoskeletal and connective tissue disorders) | 1
Pain- right flank (Musculoskeletal and connective tissue disorders) | 1
Weakness (lower extremity) (Musculoskeletal and connective tissue disorders) | 1
pain, bone (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory Loss (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Paresthesia, left foot (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 2
Personality change (Psychiatric disorders) | 1
Psych disorder, other (Psychiatric disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Brittle nails (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin, upper R leg (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash, macular (Skin and subcutaneous tissue disorders) | 1
Rash, other (facial) (Skin and subcutaneous tissue disorders) | 1
Rash- plaque like (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Sunburn (Skin and subcutaneous tissue disorders) | 1
Tooth Extraction (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes